CLINICAL TRIAL: NCT00650832
Title: A Phase II Randomized, Controlled, Partially Blinded Trial to Investigate Dose-response of TMC114/RTV in 3-class-experienced HIV-1 Infected Subjects, Followed by an Open-label Period on the Recommended Dose of TMC114/RTV.
Brief Title: TMC114-C213: A Phase II Randomized, Controlled, Partially Blinded Trial to Investigate Dose-response of TMC114/RTV in 3-class-experienced HIV-1 Infected Patients, Followed by an Open-label Period on the Recommended Dose of TMC114/RTV.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR006775
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: HIV
Keywords: HIV, anti-infectives
MeSH Terms: interventions — Darunavir

INTERVENTIONS:
Drug: TMC114; darunavir; Prezista

SUMMARY:
The purpose of this study is to determine the antiviral activity, safety and tolerability of TMC114, formulated as an oral tablet, and administered with a low dose of ritonavir

DETAILED DESCRIPTION:
This trial consists of two parts: a partially blinded dose-finding part followed by an open-label part with the recommended dose of TMC114/RTV. The dose-finding part of this trial consisted of a randomized controlled (standard of care), partially blinded, Phase II trial to determine the antiviral activity, safety and tolerability of TMC114, formulated as an oral tablet, and administered with a low dose of ritonavir. The pharmacokinetics of TMC114 are also assessed.Three hundred HIV-1 infected patients who were three-class-experienced and who were on a stable PI-containing regimen at screening for at least 8 weeks and who had plasma HIV-1 RNA > 1000 copies/mL were eligible. Three-class experience was defined as prior treatment with ³ 2 NRTIs for at least 3 months in total and ³ 1 NNRTI as part of a failing regimen. In addition, patients had to have received at least one PI for at least 3 months in the past and had to have at least 1 primary PI mutation (according to IAS definitions) at screening.As soon as all results to determine eligibility were available, and no later than 2 weeks prior to the baseline visit, the patients were randomized to one of 4 TMC114/RTV treatment groups or to a control group (standard of care). At baseline, patients changed to an investigator selected PI(s) regimen or TMC114/RTV plus optimized background regimen (OBR) consisting of NRTIs with or without T-20.In the dose-finding part of the trial, the primary objective of the trial was to evaluate the dose-response relationship in antiviral activity between the TMC114 /RTV treatment groups at 24 weeks. The recommended dose has been selected based on two joint interim analyses of this trial and of a similar trial (TMC114-C202, conducted in the United States of America, Puerto Rico, and Argentina) including approximately 150 patients in each of the two dose-finding trials (TMC114-C202 + TMC114-C213) who reached Weeks 16 and 24 or dropped out earlier. The Week 24 interim analysis included a total of 497 patients, of whom 329 had reached Week 24 or discontinued earlier. Based on the results of these two joint interim analyses, TMC114/RTV 600/100 mg b.i.d. was selected as the recommended dose for the open-label part of this trial and for future trials in treatment-experienced HIV-1 infected patients. The recommended dose of TMC114/RTV was not communicated to the investigators until the data cut-off date for the primary efficacy analysis of the two dose-finding trials was reached.The primary efficacy analysis was performed when approximately 300 patients in this trial reached 24 weeks of treatment or discontinued earlier (i.e., the primary endpoint, which was reached on 1 February 2005; A total of 318 patients were included in the analysis of whom 301 reached Week 24 or discontinued earlier). In this primary efficacy analysis, all TMC114 groups were compared to the control group by means of the confirmed virologic response at Week 24, defined as a drop in viral load of at least 1 log10 versus baseline. This primary efficacy analysis confirmed that TMC114/RTV 600/100 mg b.i.d. is the recommended dose for treatment-experienced HIV-1 infected patients.After the primary endpoint of the trial was reached (1 February 2005), and after approval of the related protocol amendment by the relevant IEC/IRB and authorities, the patients in the TMC114/RTV groups were instructed to switch to the recommended dose of TMC114/RTV (600/100 mg b.i.d.) in the open-label part of the trial.In addition, long term safety, tolerability and the durability of antiviral activity of TMC114/RTV over 144 weeks in 3-class-experienced HIV-1 infected patients will be evaluated. The trial includes a screening period of a maximum of 6 weeks, and a 144-week treatment period followed by a 4-week follow-up period. The maximum duration of the trial will be 154 weeks.Tibotec will provide follow-up treatment with TMC114/RTV for all patients who continue to benefit from treatment with TMC114/RTV. TMC114 will be provided until the drug is commercially available or until its development is discontinued.The patient will remain on the study until he/she no longer benefits from TMC114/RTV, as judged by the investigator, or he/she meets one of the withdrawal criteria. Dose-finding part of the trial: 400 mg/100 mg q.d. TMC114/RTV or 800 mg/100 mg q.d. TMC114/RTV or 400 mg/100 mg b.i.d. TMC114/RTV or 600 mg/100 mg b.i.d. TMC114/RTV. Open-label part of the trial: 600 mg/100 mg b.i.d. TMC114/RTV. Total treatment duration of 144 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented HIV-1 infection
* Patients receiving a PI-containing regimen at screening initiated at least 8 weeks prior to screening with plasma HIV-1 RNA > 1000 copies/mL
* Prior use of more than 1 NRTI for at least 3 months in total
* Prior use of one or more NNRTIs (investigational included) as part of a failing regimen
* Patients having at least 1 primary PI mutation at screening as defined by the IAS guidelines (D30N, M46I/L, G48V, I50V/L, V82A/F/T/S, I84V, L90M)16
* patients experienced to at least one PI for a total period of at least 3 months
* Patients voluntarily signs the informed consent form
* Patients can comply with the protocol requirements
* Patients having a general medical condition that, in the investigator's opinion, does not interfere with the assessments and the completion of the trial.

Exclusion Criteria:

* Presence of any currently active AIDS defining illness with the following exceptions, which must be discussed with the sponsor prior to enrollment: Stable cutaneous Kaposi's Sarcoma (i.e. no pulmonary or gastrointestinal involvement other than oral lesions) that is unlikely to require any form of systemic therapy during the trial. Wasting syndrome due to HIV infection if, in the investigator's opinion, it is not actively progressive and its treatment does not require hospitalization or compromise the patient's safety or compliance to adhere to the study protocol procedures. If patients are on maintenance therapy (which may include human Growth Hormone, appetite stimulants and anabolic steroids) for previously diagnosed wasting, they may be eligible for the trial only if such treatment is not included in the list of disallowed medications
* Current or past history of alcohol and/or drug use which, in the investigator's opinion, would compromise the patient's safety or compliance to the study protocol procedures
* patients on a treatment interruption at screening
* patients for whom an investigational ARV is part of the regimen at screening, (with the following exceptions: T-20, FTC, atazanavir and fos-amprenavir) or use of any other non-ARV investigational agents at least 90 days prior to screening
* Use of disallowed concomitant therapy
* Previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication (TMC114/RTV/placebo)
* Life expectancy of less than 6 months
* Pregnant or breast feeding
* Female patient of childbearing potential without use of effective non-hormonal birth control methods or not willing to continue practicing these birth control methods from screening until at least 14 days after the end of the treatment period
* Patients with clinical or laboratory evidence of active liver disease, liver impairment/dysfunction or cirrhosis irrespective of liver enzyme levels
* Any active or unstable medical condition (e.g. TB
* cardiac dysfunction
* acute viral infections) or findings during screening of medical history or physical examination that, in the investigator's opinion, would compromise the patients safety or outcome of the study
* Patients with the following laboratory abnormalities as defined by ACTG grading scheme Renal impairment: serum creatinine grade 2 or greater (> 1.5 x ULN)
* Lipase grade 2 or greater (> 1.5 x ULN)
* Hemoglobin toxicity grade 2 or greater (£ 7.9 g/dL)
* Platelet count grade 2 or greater (< 75000/mm³)
* Absolute neutrophil count grade 2 or greater (£ 999/mm3)
* ALT, AST grade 2 or greater (>2.5 x ULN)
* Total bilirubin grade 2 or greater (> 1.5 x ULN) unless clinical assessment foresees an immediate health risk to the patient. For patients receiving indinavir or atazanavir at screening the total bilirubin may not exceed 3 x ULN
* Any grade 3 or 4 toxicity with the following exceptions unless clinical assessment foresees an immediate health risk to the patient: Patients with pre-existing diabetes or assessments under non-fasted conditions who experienced a glucose grade 3 or 4, Patients with triglyceride or cholesterol elevation of grade 3 or 4 under non-fasted conditions, Patients who experienced asymptomatic triglyceride or cholesterol elevations of grade 3 or 4, patients who experienced an asymptomatic and isolated GGT grade 3 or 4 elevation with all other LFTs and bilirubin within normal ranges
* Patients who have been randomized to a TMC114 treatment arm in a previous TMC114 trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2003-10; Primary Completion 2005-02 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of the trial is to compare all TMC114/RTV dose groups with control at Week 24 (the primary endpoint) by means of the confirmed virologic response, defined as a drop in viral load of at least 1 log10 versus baseline.

SECONDARY OUTCOMES:
To evaluate safety and tolerability over 24 to 144 weeks; To evaluate the durability of the antiviral activity; To investigate the dose-response by comparing the different TMC114/RTV dosages.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Result] Clotet B, Bellos N, Molina JM, Cooper D, Goffard JC, Lazzarin A, Wohrmann A, Katlama C, Wilkin T, Haubrich R, Cohen C, Farthing C, Jayaweera D, Markowitz M, Ruane P, Spinosa-Guzman S, Lefebvre E; POWER 1 and 2 study groups. Efficacy and safety of darunavir-ritonavir at week 48 in treatment-experienced patients with HIV-1 infection in POWER 1 and 2: a pooled subgroup analysis of data from two randomised trials. Lancet. 2007 Apr 7;369(9568):1169-78. doi: 10.1016/S0140-6736(07)60497-8. PMID 17416261